CLINICAL TRIAL: NCT01554657
Title: Five Versus Seven Day Antibiotic Course for the Treatment of Pneumonia in the Intensive Care Unit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201108280
Record Dates: First submitted 2012-03-07; First posted 2012-03-15 (Estimated); Last update posted 2012-03-15 (Estimated); Status verified 2012-03

CONDITIONS: Pneumonia, Bacterial
Keywords: Pneumonia, Bacterial
MeSH Terms: conditions — Pneumonia, Bacterial | interventions — Anti-Bacterial Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 5 Days (Experimental)
  Interventions: Other: 5 Days of Antibiotics
- 7 days (Placebo Comparator)
  Interventions: Other: 7 Days of Antibiotics therapy for pneumonia

INTERVENTIONS:
Other: 5 Days of Antibiotics — The choice of the specific antibiotic is made by the treating intensive care unit attending physician. The patients will be randomized to two separate groups based on length of antibiotic therapy not specific antibiotics. Therefore, the actual antibiotic that will be given is not determined by the study. The patients all will receive antibiotics for pneumonia chosen by the intensive care unit team, and those in this group receive a goal of 5 days.
  Arms: 5 Days
Other: 7 Days of Antibiotics therapy for pneumonia — The choice of the specific antibiotic is made by the treating intensive care unit attending physician. The patients will be randomized to two separate groups based on length of antibiotic therapy not specific antibiotics. Therefore, the actual antibiotic that will be given is not determined by the study. The patients all will receive antibiotics for pneumonia that is determined by the treating intensive care unit team, and those in this group receive a goal of 7 days.
  Arms: 7 days

SUMMARY:
The goal of the study is to determine if patients who are being treated for pneumonia in the intensive care unit can be safely treated with five days of antibiotics (the current standard is seven to eight days). The goal is to determine if the investigators can minimize antibiotic complications while still treating the infection. Patients in the study are randomly assigned to either receive antibiotics for a goal of five days or a goal of seven days. Every patient is followed daily, and if they are not responding to the antibiotics, the treating team in the intensive care unit care can continue the antibiotics for a longer course regardless of what group the patient is assigned. The investigator's hypothesis is that patients in the five day treatment goal will be able to receive less antibiotics than patients in the seven day treatment goal without any adverse effects.

DETAILED DESCRIPTION:
This is a pilot study to determine if patients with pneumonia in the intensive care unit can safely receive five days of antibiotics. All patients admitted to the medical and surgical intensive care units at Barnes-Jewish Hospital with pneumonia will be screened for the inclusion and exclusion criteria. Patients will be randomized by sealed envelopes in groups of six to a five or seven day course of antibiotics. The choice of the antibiotic to be used is determined by the intensive care unit treating team. The patients will NOT be randomized to a specific antibiotic. The patients will be followed for a clinical response by improvement in maximum daily temperature, white blood cell count, and PaO2 to FiO2 ratio. Antibiotics can continue past the goal duration for patients in either group if the above criteria are not met or if the attending physician in the intensive care unit feels that a longer course is needed. The treating team in the intensive care unit will not be blinded to the patient's treatment assignment.

ELIGIBILITY:
Inclusion Criteria:

* New diagnosis of pneumonia
* Patient in medical or surgical intensive care unit
* Age greater or equal than 18 years old

Exclusion Criteria:

* Neutropenia
* Recipient of a solid organ or bone marrow transplant
* Bacteremia
* Presence of Acinetobacter baumannii or Stenotrophomonas maltophilia from a respiratory tract culture
* Presence of a second infection requiring antibiotic therapy
* Pregnancy
* Enrollment in another clinical study
* Patient or surrogate unable to provide informed consent
* Attending intensive care unit physician declined enrollment in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2011-01; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Length of antibiotic therapy | 28 days

SECONDARY OUTCOMES:
Mortality | 28 days
Hospital Length of Stay | 28 Days
Clostridium difficile diarrhea | 28 Days
Development of a new multi-drug resistant bacteria from a lower respiratory tract culture | 28 days
  Patients will not receive routine follow-up respiratory cultures as part of the protocol. However, if a culture is obtained on a clinical basis and the culture grows a new multi-drug resistant bacteria, then this outcome is met. The outcome does NOT have a specific unit of measure as it is a measure of whether a multi-drug resistant bacteria is present or not. The definition for a multi-drug resistant bacteria is based on the definition provided by the European Centers for Disease Control.
Recurrent lower respiratory tract infection | 28 days